CLINICAL TRIAL: NCT00122187
Title: Translation of Colorectal Cancer Screening Guidelines: A System Intervention
Brief Title: Translation of Colorectal Cancer Screening Guidelines to Practice: A System Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRT 02-059
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: cancer; colonoscopy; mass screening; colorectal cancer; colorectal carcinoma; reminder systems; rectal cancers; colorectal tumor; guidelines; CRC secondary prevention; colorectal neoplasms; colonic neoplasms; colonic diseases; hemoccult testing
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Consult System (Experimental): A new consult system designed to automatically send a gastroenterology consult request for patients with positive fecal occult blood testing (FOBT+) results
  Interventions: Device: Electronic Consult System
- Usual Care (No Intervention): The usual and customary procedures for addressing FOBT+ results: primary care physicians continued to be responsible for follow up of FOBT+ results.

INTERVENTIONS:
Device: Electronic Consult System — Consult system is an event notification system programmed to function within the VA electronic medical record system.
  Arms: Electronic Consult System

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer-related deaths in the United States. Results from randomized clinical trials and intervention studies have suggested that implementation of a CRC screening program for men and women over age 50 results in reduced CRC mortality. However, for this reduction to be fully realized, it is imperative that all positive screening tests are followed by complete diagnostic evaluation (CDE). Numerous intervention programs have been used to improve initial CRC screening rates, but data indicate that outside the research setting, less than half of patients with a positive fecal occult blood test (FOBT) screening result undergo CDE. To enhance the translation of this best practice recommendation to clinical practice, the investigators propose to implement an electronic event notification intervention (CRC-ENS) directed at making physician and system level changes to increase the proportion of patients with an abnormal FOBT that undergo CDE.

DETAILED DESCRIPTION:
Objectives: 1.To implement an electronic CRC screening event notification system intervention to improve complete evaluation of patients with a positive FOBT at four of eight VAMCs randomized to this intervention vs usual care.

2.To conduct a qualitative evaluation to identify implementation barriers and facilitators, and to guide modifications of the CRC-ENS. 3.To conduct an outcome evaluation to determine the effectiveness of the intervention to:

a. increase the proportion of patients with a positive FOBT receiving CDE. b. reduce the time-lag between notification of a positive FOBT result and scheduling of a follow-up endoscopic procedure. 4. To improve patient compliance with follow-up recommendations through combined scheduling.

Methods: The CRC-ENS intervention employs a relatively simple alteration to the current electronic mechanism for notifying the primary care provider (PCP) of when a positive FOBT is recorded. With the CRC-ENS, this notification will be forwarded to the gastroenterology (GI) clinic as well as the PCP. This notification at the GI clinic will set off a cascade of events that would normally only be triggered by a consult request from the PCP. In this translation study, eight participating VHA sites will be randomly assigned to either the CRC-ENS intervention or usual care group. The proposed project will take two years to complete. During the first project year, the participating sites will be recruited and randomized. Pre-intervention change of awareness strategies will be initiated at all intervention sites. The CRC-ENS intervention will be implemented in the second project year, and formative evaluation (including two sets of focus groups) will be carried out throughout the intervention period. Post-intervention data collection, outcome evaluation and dissemination of results will be carried out in months 18-24.

ELIGIBILITY:
Inclusion Criteria:

- VA Medical Centers with either CORI (Clinical Outcomes Research Initiative) or electronic notes/descriptions documenting GI endoscopic procedures

Exclusion Criteria:

- VA Medical Centers without electronic GI procedure documentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L. Humphrey, MD MPH, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (9):
- United States (9):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - Minneapolis, Minneapolis, Minnesota
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA Medical & Regional Office Center, White River, White River Junction, Vermont

REFERENCES:
- [Result] Tsai TT, Nallamothu BK, Prasad A, Saint S, Bates ER. Clinical problem-solving. A change of heart. N Engl J Med. 2009 Sep 3;361(10):1010-6. doi: 10.1056/NEJMcps0903023. No abstract available. PMID 19726776
- [Result] Messersmith WA, Ahnen DJ. Targeting EGFR in colorectal cancer. N Engl J Med. 2008 Oct 23;359(17):1834-6. doi: 10.1056/NEJMe0806778. No abstract available. PMID 18946069
- [Result] Humphrey LL, Shannon J, Partin MR, O'Malley J, Chen Z, Helfand M. Improving the follow-up of positive hemoccult screening tests: an electronic intervention. J Gen Intern Med. 2011 Jul;26(7):691-7. doi: 10.1007/s11606-011-1639-3. Epub 2011 Feb 15. PMID 21327529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 8 Veterans Affairs medical centers (VAMCs) to be involved with this trial evaluating a new method of processing positive colorectal cancer screening tests compared with usual care. 4 VAMCs (2 control and 2 intervention sites) dropped out of the study and 4 completed it.
Pre-assignment Details: Participating VAMCs were chosen that had electronic registries for gastroenterology (GI) endoscopic procedures available.
Period: Overall Study
Arm/Group | Electronic Consult System | Usual Care
Started | 4 | 4
Matched by Colonoscopy Volume | 4 | 4
Randomized to Intervention or Usual Care | 4 | 4
Intervention Implemented | 3 | 4
Post-intervention Data Collection | 2 | 2
Completed | 2 | 2
Not Completed | 2 | 2
Not completed — Withdrew because of resource limitations | 2 | 2

BASELINE CHARACTERISTICS:
Population: The population is the number of VAMCs that enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Electronic Consult System | Usual Care | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Customized [Number; unit: participants] — Participants in this study were VAMCs rather than human subjects. Age of participants was not collected because it was not applicable.
  participants
    Not collected | 4 | 4 | 8
Sex/Gender, Customized [Number; unit: participants] — Participants in this study were VAMCs rather than human subjects. Gender of participants was not collected because it was not applicable.
  participants
    Not collected | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Receiving GI Consult for FOBT+ Results
Description: Percent of patients receiving GI consult within 30, 90, and 180 days of FOBT+ results
Time Frame: 6 months
Population: Sites that completed the intervention and post-intervention data collection were included in the analysis
Measure: Number; unit: percent patients receiving GI consult
Groups:
- Electronic Consult System 1st Site (1a): A new consult system designed to automatically send a gastroenterology consult request for patients with positive fecal occult blood testing (FOBT+) results
- Electronic Consult System 2nd Site (2a): A new consult system designed to automatically send a gastroenterology consult request for patients with FOBT+ results
- Usual Care 1st Site (1b); Usual Care 2nd Site (2b): The usual and customary procedures for addressing FOBT+ results: primary care physicians continued to be responsible for follow up of FOBT+ results.
Arm/Group | Electronic Consult System 1st Site (1a) | Electronic Consult System 2nd Site (2a) | Usual Care 1st Site (1b) | Usual Care 2nd Site (2b)
Number analyzed (Participants) | 1 | 1 | 1 | 1
percent patients receiving GI consult
  pre intervention--consult within 30 days FOBT+ | 39 | 47 | 64 | 51
  post intervention--consult within 30 days FOBT+ | 68 | 80 | 63 | 48
  pre intervention--consult within 90 days FOBT+ | 46 | 50 | 70 | 56
  post intervention--consult within 90 days FOBT+ | 72 | 82 | 69 | 56
  pre intervention--consult within 180 days FOBT+ | 50 | 55 | 71 | 62
  post intervention--consult within 180 days FOBT+ | 74 | 86 | 72 | 59

2. Primary Outcome: Percent of Patients Receiving GI Consult Plus Anatomic Workup for FOBT+ Results
Description: Percent of patients receiving GI consult plus anatomic workup within 30, 90, and 180 days of FOBT+ results
Time Frame: 6 months
Population: Sites that completed the intervention and post-intervention data collection were included in the analysis
Measure: Number; unit: percent patients with GI consult+workup
Arm/Group | Electronic Consult System 1st Site (1a) | Electronic Consult System 2nd Site (2a) | Usual Care 1st Site (1b) | Usual Care 2nd Site (2b)
Number analyzed (Participants) | 1 | 1 | 1 | 1
percent patients with GI consult+workup
  pre intervention--consult+workup in 30 days FOBT+ | 4 | 12 | 19 | 4
  post intervention--consult+workup in 30 days FOBT+ | 30 | 21 | 13 | 5
  pre intervention--consult+workup in 90 days FOBT+ | 18 | 26 | 44 | 15
  post intervention--consult+workup in 90 days FOBT+ | 49 | 39 | 50 | 17
  pre intervention--consult+workup in 180days FOBT+ | 25 | 29 | 48 | 22
  post intervention--consult+workup in 180days FOBT+ | 51 | 42 | 54 | 22

ADVERSE EVENTS:
Description: Adverse events were not formally monitored because participants were VAMCs, not human subjects. The study involved extracting information from individual medical records at each VAMC. There were no reported problems involving this use of records.
Arm/Group | Electronic Consult System | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Half of the sites randomized did not complete the study. GI referral rates should have been nearly 100%, yet were not. Because of programming limitations, we were unable to evaluate the type of diagnostic interventions the patients received.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes